CLINICAL TRIAL: NCT03576573
Title: Post Market Clinical Follow-Up Study Protocol for PROCOTYL® C Acetabular Components
Status: Enrolling by invitation | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002N
Record Dates: First submitted 2018-06-26; First posted 2018-07-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Joint Disease
Keywords: Osteoarthritis; Avascular necrosis; Ankylosis; Protrusio acetabuli; Painful hip dysplasia; Rheumatoid arthritis; Correction of functional deformity
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Total Hip Arthroplasty: Single arm study of subjects previously implanted with any MicroPort Orthopedics or Wright Medical Technology femoral stems and PROCOTYL® C Acetabular Components
  Interventions: Device: PROCOTYL® C

INTERVENTIONS:
Device: PROCOTYL® C — Hip Arthroplasty
  Other Names: Primary Total Hip Device

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) components marketed in the European Union (EU). These types of studies are required by regulatory authorities for all THA devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in Europe. This study has been designed in accordance with the medial device directives (MEDDEV) 2.12/2 rev 2.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, subjects must meet all of the following criteria:

* Has previously undergone primary Total Hip Arthroscopy for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;
* Inflammatory degenerative joint disease such as rheumatoid arthritis;
* Correction of functional deformity
* Subject was implanted with the specified combination of components, namely, any MicroPort Orthopedics or Wright Medical Technology femoral stem and PROCOTYL C Acetabular Components
* Subject is willing and able to complete required study visits or assessments

Previously implanted bilateral subjects can have both THAs (Total Hip Arthroscopy) enrolled in the study provided:

1. the specified combination of components were implanted in both,
2. all other aspects of the Inclusion/Exclusion Criteria are satisfied,
3. enrollment does not exceed the subject count specified in the Clinical Trial Agreement, and
4. the subject agrees to a second Informed Consent document specific to the second THA. Prospective enrolment of a previously unimplanted hip is not permitted in this study.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* Subject was skeletally immature (less than 21 years of age) at time of implantation
* Subject has a non-MicroPort or non-Wright Medical Technology component implanted (femoral heads, acetabular shells, acetabular liners) in the enrolled Total Hip Arthroscopy
* Subject is currently enrolled in another clinical investigation which could affect the endpoints of this protocol
* Subject is unwilling or unable to sign the Informed Consent document
* Subject has documented substance abuse issues
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
* Subject is currently incarcerated or has impending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously implanted with any MicroPort Orthopedics or Wright Medical Technology Femoral Stems and PROCOTYL® C Acetabular Components
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary endpoint is to evaluate component survivorship of the PROCOTYL® C Acetabular Components out to 10 years follow-up. Percentage of hips survived with no revision or replacement at 10-year.

SECONDARY OUTCOMES:
To determine the cumulative incidence of component revision at specified intervals out to 10 years follow-up; | 2-5 years, 5-7 years, and 10 years
  Percentage of hips that were revised or replaced at each of the intervals namely for Early (2-5 years), midterm (5-7 Year), and long-term (10-year) evaluation.
To characterize functional scores, as assessed by Oxford Hip. | 2-5 years, 5-7 years, and 10 years
  The study will be reporting the final Oxford Hip score, which is a summary over 12 items. Each of these items is 5-level Likert scale such as from 'not at all' to 'totally'.
To characterize functional scores, as assessed by EQ-5D-3L scores. | 2-5 years, 5-7 years, and 10 years
  EQ-5D-3L data will be summarized over 5 domains, namely, mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain has 3 levels: no problems, some problems, and extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Elbe Kliniken Buxtehude, Buxtehude, Germany

IPD SHARING:
Plan to Share IPD: No